CLINICAL TRIAL: NCT02422953
Title: Effectiveness of Food/Nutrient Based Interventions to Prevent Stunting Among Children Under Five in Thatta and Sujawal Districts, Sindh Province, Pakistan
Brief Title: Stunting Prevention Project in Thatta and Sujawal Districts, Sindh Province, Pakistan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: United Nations World Food Programme (WFP) (Other); Pakistan Ministry of Health (Other Government)
Responsible Party: Principal Investigator, Dr Sajid Bashir Soofi, Associate Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WFP-Thatta
Record Dates: First submitted 2015-04-15; First posted 2015-04-22 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Malnutrition
Keywords: Stunting; Wasting; Underweight
MeSH Terms: conditions — Malnutrition; Growth Disorders; Cachexia; Thinness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Wheat Soya Blend, Wawa Mum, Micronutrient Powders, Behavior change and preventive health massages
  Interventions: Dietary Supplement: Wheat Soya Blend (WSB); Dietary Supplement: Wawa Mum; Dietary Supplement: Micronutrient Powders (MNP); Behavioral: Behavior change and preventive health massages
- Control (No Intervention): Control group will receive routine public and private health services available in the area.

INTERVENTIONS:
Dietary Supplement: Wheat Soya Blend (WSB) — A monthly ration of 5 Kg of Wheat Soya Blend (WSB) will be given to pregnant women every month during pregnancy and lactating mothers for six months after giving birth
  Arms: Intervention
Dietary Supplement: Wawa Mum — Children 6-23 months of age will receive a daily ration of 50 gram of Wawa Mum during study period
  Arms: Intervention
Dietary Supplement: Micronutrient Powders (MNP) — Children 24-59 months of age will receive a sachet of Micronutrient Powders (MNP) in alternate days
  Arms: Intervention
Behavioral: Behavior change and preventive health massages — Behavior change and preventive health massages will be delivered by lady health workers (LHWs) during monthly visits and in group meetings
  Arms: Intervention

SUMMARY:
Widespread food insecurity and malnutrition are largely the main impairing factors for human capital development in Pakistan. Rates of chronic malnutrition are very high, and acute malnutrition is critical: 44% of children under five are stunted and nationwide global acute malnutrition (GAM) rates amongst children under five exceed the WHO critical threshold of 15%. Nutritional status trends also show a deteriorating situation since 1994, when stunting rates were at 36%.

This study evaluates the effectiveness of food based interventions to prevent stunting among children under-five years with focus on window of opportunity (1000 days from conception to 2 years) for addressing stunting. Pregnant women, lactating mothers and children 6-59 months will receive supplements on monthly basis in intervention areas, while participants in control areas will receive routine public health services available in the study area.

DETAILED DESCRIPTION:
Children under two are consuming less than half of their daily energy requirements (560 kcal) and lower than recommended levels of micronutrients (one-third of reference nutrient intake for Iron and one-half for Zinc). Overall, less than 4% of children were receiving an acceptable, diverse diet. Food security and nutrition situation in Sindh province is even more dramatic. According to the National Nutrition Survey, 2011, GAM prevalence exceeds 18% while anemia levels amongst children under five reached the alarming level of 72.5%. With this high level of poverty and food insecurity, a food based approach to prevent stunting, together with non- food based approaches is needed.

Therefore, Division of Women and Child Health, Aga Khan University proposes a research study for stronger evidence base on the effectiveness of preventive food/nutrient based interventions on reduction of stunting and developing viable programmes on nutrition under "real" operational conditions. The effectiveness of the project will be measured in terms of the impact of the proposed interventions on the stunting and micronutrient deficiency prevalences in the target group (children and mothers). Given the conditions of project implementation, a quasi-experimental "double difference" design would be appropriate to assess the impact of the intervention. We propose to compare the intervention and non-intervention (control) groups before (first difference) and after the intervention (second difference). Then, the operational implementation of the research comprises a baseline and end line surveys. In addition, a nested cluster randomized controlled trial will be implemented to track the evolution of key variables related to the quality of intervention delivery and intermediate nutrition outcomes. The control clusters will receive routine public and private health services available in the area.

To achieve its purpose and objectives the project design includes core interventions such as complementary feeding using food/nutrient based supplements along with behavior change communication, complemented with other non-food interventions. Using a preventative (blanket) approach, three types of food/nutrient supplements (Wawamum, MNP & WSB) are considered as part of the interventions.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women
* All lactating mothers (upto 6 months)
* All children 6-23 months of age
* All children 24-59 months of age

Exclusion Criteria:

* Refuse to participate in the study
* Having severe chronic disease

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4020 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Stunting-reduction in stunted children in intervention group | 2 Years
  To calculate HAZ scores the 2006 WHO growth reference will be used

SECONDARY OUTCOMES:
Pregnancy out come | 2 Years
  Reduction in low birth weight in newborns
Mean change in weight-for-height z-score (WHZ) | 2 Years
  To calculate WHZ scores the 2006 WHO growth reference will be used
Mean change in weight-for-age z-score (WAZ) | 2 Years
  To calculate WAZ scores the 2006 WHO growth reference will be used
Improvement in infant and young child feeding (IYCF) indicators | 2 Years
  Monthly data collection on IYCF practices
Linear growth velocity (HAZ increment/month) | 2 Years
  To calculate HAZ score the 2006 WHO growth reference will be used
Mean hemoglobin concentration in children 6-59 months of age | 2 Years
  Hemocue will be used to measure Hb concentration
Prevalence of childhood anemia (Hb concentration<11g/dL) in children 6-59 months of age | 2 Years
  Hb spot testing will be conducted
Mean hemoglobin concentration in mothers | 2 Years
  Hemocue will be used to measure Hb concentration
Prevalence of maternal anemia (Hb concentration<12g/dL) | 2 Years
  Hb spot testing will be conducted
Impact on maternal BMI | 2 Years
  The change in BMI z-score weight and height will be combined to report BMI in kg/m^2
Impact on vitamin A status in children at 24 months | 2 Years
  The change in Vitamin A status (µmol/L) in children at 24 months of age
Impact on vitamin D status in children at 24 months | 2 Years
  The change in vitamin D status (ng/mL) in children at 24 months of age
Impact on Zinc status in children at 24 months | 2 Years
  The change in Zinc status (µg/dL) in children at 24 months of age
Impact on Ferritin status in children at 24 months | 2 Years
  The change in Ferritin status (ng/mL) in children at 24 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Sajid B Soofi, FCPS, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Data are sharing with funding agency on 6-monthly basis
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: As per the project deliverables
Access Criteria: Review and feedback
URL: https://www.wfp.org

REFERENCES:
- [Background] National Nutrition Survey (NNS), 2011. Planning Commission Planning and Development Division Government of Pakistan.
- [Background] WFP (2012): Protracted Relief and Recovery Operations (PRRO). Pakistan 200250. Rome, Italy.
- [Background] Horton, S. Opportunities for investments in nutrition in low-income Asia; 1999. Asian Development Review 17 (1, 2): 246-273.
- [Background] Gorstein J, Sullivan KM, Parvanta I, Begin F. Indicators and Methods for Cross-Sectional Surveys of Vitamin and Mineral Status of Populations. The Micronutrient Initiative (Ottawa) and the Centers for Disease Control and Prevention (Atlanta), May 2007.
- [Background] Donner, A. and Klar, N. Design and Analysis of Cluster Randomization Trials in Health Research. Arnold, London; 2000
- [Derived] Soofi SB, Khan GN, Ariff S, Ihtesham Y, Tanimoune M, Rizvi A, Sajid M, Garzon C, de Pee S, Bhutta ZA. Effectiveness of nutritional supplementation during the first 1000-days of life to reduce child undernutrition: A cluster randomized controlled trial in Pakistan. Lancet Reg Health Southeast Asia. 2022 Jul 19;4:100035. doi: 10.1016/j.lansea.2022.100035. eCollection 2022 Sep. PMID 37383995
- [Derived] Khan GN, Kureishy S, Ariff S, Rizvi A, Sajid M, Garzon C, Khan AA, de Pee S, Soofi SB, Bhutta ZA. Effect of lipid-based nutrient supplement-Medium quantity on reduction of stunting in children 6-23 months of age in Sindh, Pakistan: A cluster randomized controlled trial. PLoS One. 2020 Aug 13;15(8):e0237210. doi: 10.1371/journal.pone.0237210. eCollection 2020. PMID 32790725
- [Derived] Zaidi S, Das JK, Khan GN, Najmi R, Shah MM, Soofi SB. Food supplements to reduce stunting in Pakistan: a process evaluation of community dynamics shaping uptake. BMC Public Health. 2020 Jul 2;20(1):1046. doi: 10.1186/s12889-020-09103-8. PMID 32616009
- [Derived] Kureishy S, Khan GN, Arrif S, Ashraf K, Cespedes A, Habib MA, Hussain I, Ullah A, Turab A, Ahmed I, Zaidi S, Soofi SB. A mixed methods study to assess the effectiveness of food-based interventions to prevent stunting among children under-five years in Districts Thatta and Sujawal, Sindh Province, Pakistan: study protocol. BMC Public Health. 2017 Jan 5;17(1):24. doi: 10.1186/s12889-016-3976-y. PMID 28056945